CLINICAL TRIAL: NCT01330680
Title: Genetic Determinants of Cardiovascular Response to Coffee Drinking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: G. d'Annunzio University (Other)
Collaborators: Institute for Scientific Information on Coffee (Other); Italian Istituto Nazionale Ricerche Cardiovascolari (Unknown)
Responsible Party: Raffaele De Caterina/MD, PhD, Institute of Cardiology, G. d'Annunzio University of Chieti
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: C041003
Record Dates: First submitted 2011-03-29; First posted 2011-04-07 (Estimated); Last update posted 2011-04-07 (Estimated); Status verified 2011-03

CONDITIONS: Caffeine
Keywords: coffee; caffeine; blood pressure; nutrigenetics; gene polymorphisms; Acute Cardiovascular and Neuropsychologic Effects
MeSH Terms: interventions — Coffee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Coffee (Experimental)
  Interventions: Dietary Supplement: Coffee
- Decaffeinated coffee (Active Comparator)
  Interventions: Dietary Supplement: Decaffeinated coffee

INTERVENTIONS:
Dietary Supplement: Coffee — 40 mL dose of a decaffeinated preparation spiked with the addition of caffeine, at a dose of 3 mg/kg
  Arms: Coffee
Dietary Supplement: Decaffeinated coffee — 40 mL dose of decaffeinated coffee
  Arms: Decaffeinated coffee

SUMMARY:
Cardiovascular and neuropsychologic effects of coffee are still debated. The precise mechanism underlying the actions of caffeine on the cardiovascular and neuropsychologic systems is incompletely understood and a considerable variability in the response to coffee drinking was observed, in part ascribable to a genetic trait.

The aim of the study is to evaluate acute cardiovascular and neuropsychologic effects of coffee and explore whether such effects are influenced by the genetic asset of caffeine metabolism (by a polymorphisms of cytochrome P450 1A2), adenosine metabolism (by polymorphisms of adenosine receptor and adenosine monophosphate deaminase) or catecholamine receptors (by polymorphisms of adrenergic receptors).

DETAILED DESCRIPTION:
Coffee is among the most widely consumed beverages worldwide. Despite the relationship between coffee consumption and the incidence of cardiovascular disease has been studied extensively, the effects of this drink on the cardiovascular apparatus and its role as a risk factor for coronary heart disease are still debated. Moreover, the effect of coffee on attention, sleep changes, anxiety and panic disorders was studied but a great variability was observed.

Many of the known or suspected cardiovascular and neuropsychologic effects of coffee have been attributed to caffeine. The main mechanism of action of caffeine is to antagonize adenosine receptors; a secondary effect is the inhibition of phosphodiesterases, with the subsequent accumulation of cyclic adenosine monophosphate and a intensification of the effects of catecholamines.

It is also well known that there is a considerable variability in the cardiovascular and neuropsychologic response to coffee drinking, explaining the inconsistency between different effects observed in the various studies. This variability may have a genetic basis.

The aim of the study is to evaluate acute cardiovascular and neuropsychologic effects of coffee and explore whether such effects are influenced by the genetic asset of caffeine metabolism (by a polymorphisms of cytochrome P450 1A2), adenosine metabolism (by polymorphisms of adenosine receptor and adenosine monophosphate deaminase) or catecholamine receptors (by polymorphisms of adrenergic receptors).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 40 years
* Males (to avoid variation due to female hormonal cycle)
* No known active ongoing disease (apparent good health)
* Non-smokers (to avoid contributory effects of nicotine or other tobacco alkaloids to caffeine effects or tolerance)
* Average coffee intake (not less than one cup/day and not greater than three cups/day)

Exclusion Criteria:

* Treatment with any drug with known activity on the adrenergic system
* Hypertension
* Therapy with sympathomimetic drugs, theophylline, alpha- or beta-blockers, any antihypertensive therapy
* Body mass index (BMI) > 30 kg/m2 (obesity)
* BMI < 18.5 kg/m2

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2004-09; Primary Completion 2006-12 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Change in platelet aggregation | From baseline to 30 minutes and 2 hours after coffee or decaffeinated alternatively
  Light transmission aggregometry (LTA) induced by ADP and apinephrine. Platelet function analyzer (PFA) by collagen-ADP and collagen-epinephrine cartridges.
Change in cognitive tasks measures | From 30 minutes until 2 hours after coffee or decaffeinated alternatively
  Low intensity task of focused attention and choice reaction times (Categorical Search Task).
  More demanding response interference tasks (Letter Flanker Task). Classic interference task (Stroop Test).
Change in blood pressure | From baseline until 2 hours after coffee or decaffeinated alternatively
Change in heart rate | From baseline until 2 hours after coffee or decaffeinated alternatively

SECONDARY OUTCOMES:
Change in plasma caffeine concentration | From baseline to 30 minutes and 2 hours after coffee or decaffeinated alternatively
Change in plasma adrenaline and noradrenaline concentration | From baseline to 30 minutes and 2 hours after coffee or decaffeinated alternatively

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Cardiology - Center of Excellence on Aging, G. d'Annunzio University, Chieti, Italy

REFERENCES:
- [Background] 1) Hartley TR, Lovallo WR, Whitsett TL. Cardiovascular effects of caffeine in men and women. Am J Cardiol 2004;93:1022-6. 2) Lopez-Garcia E, van Dam RM, Willett WC, et al. Coffee consumption and coronary heart disease in men and women: a prospective cohort study. Circulation 2006;113:2045-53. 3) Silletta MG, Marfisi R, Levantesi G, et al. Coffee consumption and risk of cardiovascular events after acute myocardial infarction: results from the GISSI (Gruppo Italiano per lo Studio della Sopravvivenza nell'Infarto miocardico)-Prevenzione trial. Circulation 2007;116:2944-51. 4) Yang A, Palmer AA, de Wit H. Genetics of caffeine consumption and responses to caffeine. Psychopharmacology (Berl) 2010;211:245-57. 5) Cornelis MC, El-Sohemy A, Kabagambe EK, Campos H. Coffee, CYP1A2 genotype, and risk of myocardial infarction. JAMA 2006;295:1135-41. 6) Fredholm BB. Astra Award Lecture. Adenosine, adenosine receptors and the actions of caffeine. Pharmacol Toxicol 1995;76:93-101. 7) Anderson JL, Habashi J, Carlquist JF, et al. A common variant of the AMPD1 gene predicts improved cardiovascular survival in patients with coronary artery disease. J Am Coll Cardiol 2000;36:1248-52. 8) Snapir A, Heinonen P, Tuomainen TP, et al. An insertion/deletion polymorphism in the alpha2B-adrenergic receptor gene is a novel genetic risk factor for acute coronary events. J Am Coll Cardiol 2001;37:1516-22. 9) Bengtsson K, Melander O, Orho-Melander M, et al. Polymorphism in the beta(1)-adrenergic receptor gene and hypertension. Circulation 2001;104:187-90. 10) White HL, Maqbool A, McMahon AD, et al. An evaluation of the beta-1 adrenergic receptor Arg389Gly polymorphism in individuals at risk of coronary events. A WOSCOPS substudy. Eur Heart J 2002;23:1087-92. 11) Brodde OE. Beta-1 and beta-2 adrenoceptor polymorphisms: functional importance, impact on cardiovascular diseases and drug responses. Pharmacol Ther 2008;117:1-29.
- [Derived] Renda G, Zimarino M, Antonucci I, Tatasciore A, Ruggieri B, Bucciarelli T, Prontera T, Stuppia L, De Caterina R. Genetic determinants of blood pressure responses to caffeine drinking. Am J Clin Nutr. 2012 Jan;95(1):241-8. doi: 10.3945/ajcn.111.018267. Epub 2011 Dec 14. PMID 22170367